CLINICAL TRIAL: NCT05325021
Title: Correction of Anisometropic Amblyopia in Children at School Age.
Brief Title: Correction of Anisometropic Amblyopia in Children.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Other Study IDs: RC 7-22
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Amblyopia; Anisometropic Amblyopia; Anisometropia and Aniseikonia; Refractive Errors
Keywords: amblyopia; axial refractive error; anisometropia
MeSH Terms: conditions — Amblyopia; Anisometropia; Aniseikonia; Refractive Errors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Axial myopia: children have anisometropia due to axial myopia, axial length will be measured by optical biometry device in millimeter (mm).
  Interventions: Diagnostic Test: Axial length measurement in millimeter (mm) by optical biometry device; Diagnostic Test: Autorefractometer to measure the refractive error in both eyes.
- Refractive myopia: children have anisometropia due to refractive myopia, axial length will be measured by optical biometry device in mm.
  Interventions: Diagnostic Test: Axial length measurement in millimeter (mm) by optical biometry device; Diagnostic Test: Autorefractometer to measure the refractive error in both eyes.
- Axial hyperopia: children have anisometropia due to axial hyperopia, axial length will be measured by optical biometry device in mm.
  Interventions: Diagnostic Test: Axial length measurement in millimeter (mm) by optical biometry device; Diagnostic Test: Autorefractometer to measure the refractive error in both eyes.
- Refractive hyperopia: children have anisometropia due to refractive hyperopia, axial length will be measured by optical biometry device in mm.
  Interventions: Diagnostic Test: Axial length measurement in millimeter (mm) by optical biometry device; Diagnostic Test: Autorefractometer to measure the refractive error in both eyes.

INTERVENTIONS:
Diagnostic Test: Axial length measurement in millimeter (mm) by optical biometry device — Axial length measurement of the anisometropic eye and the fellow one in millimeter (mm) by optical biometry device.
Diagnostic Test: Autorefractometer to measure the refractive error in both eyes. — Measurement of the refractive state of both eyes for each subject to asses the refractive error in diopter (D).

SUMMARY:
Anisometropic amblyopia among children in school age may affects quality of life and educational progress of children.

DETAILED DESCRIPTION:
Correction of anisometropic amblyopia depends on type of refractive error and axial length of the eye.

In this study, we will asses the types of anisometropia found in children at school age and investigate possible ways for correction of this type of amblyopia.

ELIGIBILITY:
Inclusion Criteria:

* Anisometropic amblyopia.
* Children at school age ranged from 4 to 12 years old.

Exclusion Criteria:

* Emmetropia children.
* Children had undergone any intraocular surgeries.
* Other types of amblyopia.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Residents of a Banha city that were diagnosed as anisometropic amblyopia and are seeking refractive error corrections.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Axial length of both eyes. | Immediately after optical biometry test for each eye.
  Measurement of axial length of both eyes in millimeter (mm).

SECONDARY OUTCOMES:
Incidence of refractive errors in anisometropic amblyopia | Immediately after autorefractometer test for each eye.
  Type of refractive error found in anisometropia measured by autorefractometer in diopter (D).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tabl, MD, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy Tabl, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Undecided